CLINICAL TRIAL: NCT00910390
Title: Randomized Comparison to Freeze Human Embryos by Either Vitrification or Slow Freezing Protocols
Brief Title: Comparison Between Three Freezing Protocols to Preserve Human Embryos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Fasano Giovanna, Clinical Embryologist, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VITR-1-EMBRYOS
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2016-07-26 (Estimated); Status verified 2016-07

CONDITIONS: Human Embryo Cryopreservation
Keywords: IVF; embryo cryopreservation; vitrification; Human Embryo; Embryonic development; Pregnancy rate
MeSH Terms: interventions — Propylene Glycol; Ethylene Glycol; Dimethyl Sulfoxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Slow Freezing (Placebo Comparator): Standard freezing protocol (slow freezing) of preimplantation embryos
  Interventions: Other: Slow freezing
- VIT-Irvine (Experimental): Vitrification with Irvine solution (rapid freezing) of preimplantation embryos
  Interventions: Other: VIT-Irvine
- VIT-Vitrolife (Experimental): Vitrification (rapid freezing) with Vitrolife solution
  Interventions: Other: Vit-Vitrolife

INTERVENTIONS:
Other: Slow freezing — Embryos at different developmental stages will be frozen using a solution that contains propanediol and sucrose, individually placed in high security straws, cooled with a programmator and stored in liquid nitrogen.
  Other Names: Home-made solutions; propanediol
  Arms: Slow Freezing
Other: VIT-Irvine — Embryos at different developmental stages will be frozen using the vitrification solution according to the manufacturer's instructions, individually placed in high security vitrification devices and plunged directly in liquid nitrogen for storing.
  Other Names: IRVINE, California; ethylene glycol; DMSO
  Arms: VIT-Irvine
Other: Vit-Vitrolife — Embryos at different developmental stages will be frozen using the vitrification solution according to the manufacturer's instructions, individually placed in high security vitrification devices and plunged directly in liquid nitrogen for storing.
  Other Names: VITROLIFE, Sweden; ethylene glycol; propanediol
  Arms: VIT-Vitrolife

SUMMARY:
This randomized study compares three different freezing methods to store human in vitro fertilization (IVF) embryos: vitrification with two commercial kits or slow freezing. After information, all patients undergoing IVF treatment can be included in the study. If qualified, embryos at different developmental stages will be allocated between the three methods. At the end of the first year survival and developmental rates, and implantation and pregnancy rates will be analyzed in order to determine the best method.

DETAILED DESCRIPTION:
Despite all the advances achieved in vitro fertilized treatments, it is known that the chances of implantation for fertilised in vitro embryo remain limited, at around 20%. Cryopreservation of supernumerary embryos produced during IVF cycles provides an opportunity for patients to increase the number of transfers per oocyte harvest cycle, increasing then their chances of conception.

The freezing technique may involve different media and methods, which lead to different survival and developmental rates after thawing.

Vitrification is a new freezing method, which consists in exposing cells to high concentrations of cryoprotectants and then cooling them ultra-rapidly; this induces an increase in viscosity which favours the formation of a vitreous state without any ice crystals formation. This method contrasts with the slow freezing method (currently employed), which is based on exposure to very low concentrations of cryoprotectants combined with long cooling times and associated with a higher risk of ice crystal formation.

Both methods can reduce cell survival and embryo ability to develop, either by the high concentrations of cryoprotectants in case of vitrification, or by ice crystals formation in case of slow freezing. The advantages of vitrification in embryology may be considerable because embryos seem more sensitive to ice crystal formation than to cyroportectant concentration; consequently, the elimination of office crystal injury may increase their survival chances. Additionally in the case of vitrification, the time required for equilibration and cooling is considerably reduced as well as the need for expensive equipment such as programmable machine is eliminated.

At present, vitrification and slow freezing are used for the cryopreservation of oocytes and embryos at all stages of development. Encouraging results have been obtained with vitrification, but no study has randomly compared in one study, the two protocols and cryoprotectors. The purpose of this clinic randomised study is to compare three treatments: traditional slow freezing method currently employed (control group) and two different commercial vitrification methods (experimental groups) to assess the efficacy that this technique may involve.

ELIGIBILITY:
Inclusion Criteria:

* Infertility requiring IVF

Exclusion Criteria:

* Women's age > 43 years
* Patients positive for hepatitis B or C
* Patients positive for HIV

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 584 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Survival embryo rate | one year

SECONDARY OUTCOMES:
Delivery rate | one year

CONTACTS AND LOCATIONS:
Overall Officials: Anne Delbaere, Ph.D., Study Director — Fertility Clinic, Hospital Erasme
Locations (1):
- IVF laboratory, Hospital Erasme, Route de Lennik 808, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Al-Hasani S, Ozmen B, Koutlaki N, Schoepper B, Diedrich K, Schultze-Mosgau A. Three years of routine vitrification of human zygotes: is it still fair to advocate slow-rate freezing? Reprod Biomed Online. 2007 Mar;14(3):288-93. doi: 10.1016/s1472-6483(10)60869-3. PMID 17359578
- [Background] Balaban B, Urman B, Ata B, Isiklar A, Larman MG, Hamilton R, Gardner DK. A randomized controlled study of human Day 3 embryo cryopreservation by slow freezing or vitrification: vitrification is associated with higher survival, metabolism and blastocyst formation. Hum Reprod. 2008 Sep;23(9):1976-82. doi: 10.1093/humrep/den222. Epub 2008 Jun 10. PMID 18544577
- [Background] Desai N, Blackmon H, Szeptycki J, Goldfarb J. Cryoloop vitrification of human day 3 cleavage-stage embryos: post-vitrification development, pregnancy outcomes and live births. Reprod Biomed Online. 2007 Feb;14(2):208-13. doi: 10.1016/s1472-6483(10)60789-4. PMID 17298725
- [Background] Escriba MJ, Zulategui JF, Galan A, Mercader A, Remohi J, de los Santos MJ. Vitrification of preimplantation genetically diagnosed human blastocysts and its contribution to the cumulative ongoing pregnancy rate per cycle by using a closed device. Fertil Steril. 2008 Apr;89(4):840-6. doi: 10.1016/j.fertnstert.2007.04.035. Epub 2007 Aug 6. PMID 17681342
- [Background] Huang CC, Lee TH, Chen SU, Chen HH, Cheng TC, Liu CH, Yang YS, Lee MS. Successful pregnancy following blastocyst cryopreservation using super-cooling ultra-rapid vitrification. Hum Reprod. 2005 Jan;20(1):122-8. doi: 10.1093/humrep/deh540. Epub 2004 Oct 7. PMID 15471932
- [Background] Kasai M, Mukaida T. Cryopreservation of animal and human embryos by vitrification. Reprod Biomed Online. 2004 Aug;9(2):164-70. doi: 10.1016/s1472-6483(10)62125-6. PMID 15333245
- [Background] Kattera S, Chen C. Cryopreservation of embryos by vitrification: current development. Int Surg. 2006 Sep-Oct;91(5 Suppl):S55-62. PMID 17436605
- [Background] Kuwayama M, Vajta G, Ieda S, Kato O. Comparison of open and closed methods for vitrification of human embryos and the elimination of potential contamination. Reprod Biomed Online. 2005 Nov;11(5):608-14. doi: 10.1016/s1472-6483(10)61169-8. PMID 16409712
- [Background] Kuwayama M. Highly efficient vitrification for cryopreservation of human oocytes and embryos: the Cryotop method. Theriogenology. 2007 Jan 1;67(1):73-80. doi: 10.1016/j.theriogenology.2006.09.014. Epub 2006 Oct 20. PMID 17055564
- [Background] Liebermann J, Nawroth F, Isachenko V, Isachenko E, Rahimi G, Tucker MJ. Potential importance of vitrification in reproductive medicine. Biol Reprod. 2002 Dec;67(6):1671-80. doi: 10.1095/biolreprod.102.006833. PMID 12444040
- [Background] Liebermann J, Dietl J, Vanderzwalmen P, Tucker MJ. Recent developments in human oocyte, embryo and blastocyst vitrification: where are we now? Reprod Biomed Online. 2003 Dec;7(6):623-33. doi: 10.1016/s1472-6483(10)62084-6. PMID 14748959
- [Background] Liebermann J, Tucker MJ. Comparison of vitrification and conventional cryopreservation of day 5 and day 6 blastocysts during clinical application. Fertil Steril. 2006 Jul;86(1):20-6. doi: 10.1016/j.fertnstert.2006.01.029. Epub 2006 Jun 8. PMID 16762345
- [Background] Loutradi KE, Kolibianakis EM, Venetis CA, Papanikolaou EG, Pados G, Bontis I, Tarlatzis BC. Cryopreservation of human embryos by vitrification or slow freezing: a systematic review and meta-analysis. Fertil Steril. 2008 Jul;90(1):186-93. doi: 10.1016/j.fertnstert.2007.06.010. Epub 2007 Nov 5. PMID 17980870
- [Background] Nawroth F, Rahimi G, Isachenko E, Isachenko V, Liebermann M, Tucker MJ, Liebermann J. Cryopreservation in assisted reproductive technology: new trends. Semin Reprod Med. 2005 Nov;23(4):325-35. doi: 10.1055/s-2005-923390. PMID 16317621
- [Background] Rama Raju GA, Haranath GB, Krishna KM, Prakash GJ, Madan K. Vitrification of human 8-cell embryos, a modified protocol for better pregnancy rates. Reprod Biomed Online. 2005 Oct;11(4):434-7. doi: 10.1016/s1472-6483(10)61135-2. PMID 16274602
- [Background] Stehlik E, Stehlik J, Katayama KP, Kuwayama M, Jambor V, Brohammer R, Kato O. Vitrification demonstrates significant improvement versus slow freezing of human blastocysts. Reprod Biomed Online. 2005 Jul;11(1):53-7. doi: 10.1016/s1472-6483(10)61298-9. PMID 16102287
- [Background] Takahashi K, Mukaida T, Goto T, Oka C. Perinatal outcome of blastocyst transfer with vitrification using cryoloop: a 4-year follow-up study. Fertil Steril. 2005 Jul;84(1):88-92. doi: 10.1016/j.fertnstert.2004.12.051. PMID 16009162
- [Background] Vajta G, Nagy ZP. Are programmable freezers still needed in the embryo laboratory? Review on vitrification. Reprod Biomed Online. 2006 Jun;12(6):779-96. doi: 10.1016/s1472-6483(10)61091-7. PMID 16792858
- [Background] Youssry M, Ozmen B, Zohni K, Diedrich K, Al-Hasani S. Current aspects of blastocyst cryopreservation. Reprod Biomed Online. 2008 Feb;16(2):311-20. doi: 10.1016/s1472-6483(10)60591-3. PMID 18284893